CLINICAL TRIAL: NCT01679093
Title: Antagonism Research Between Antiemetics Agents (Droperidol, Dexametasone, Ondansetron) and Acetaminophen in Thyroidectomy's Post-operative Analgesia.
Brief Title: Antagonism Research Between Antiemetics Agents and Acetaminophen in Thyroidectomy's Post-operative Analgesia.
Acronym: ANPATHY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-002701-40
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Interaction Between Antiemetic Drugs and Paracetamol
Keywords: postoperative analgesia; paracetamol; 5-HT3 antagonist; ondansetron; PainMatcher
MeSH Terms: interventions — Ondansetron; Droperidol; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ONDANSETRON (OS) (Active Comparator): patients receiving ondansetron at the beginning of the surgery to prevent postoperative nausea and vomiting (PONV); and paracetamol at the end of the surgery for postoperative analgesia.
  Interventions: Drug: ondansetron
- DROPERIDOL (DRO) (Active Comparator): patients receiving droperidol at the beginning of the surgery to prevent PONV; and paracetamol at the end of the surgey for postoperative analgesia.
  Interventions: Drug: Droperidol
- DEXAMETHASONE (DEXA) (Active Comparator): patients receiving dexamethasone at the beginning of the surgery to prevent PONV; and paracetamol at the end of the surgey for postoperative analgesia.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: ondansetron — ondansetron: 4 mg intravenous administration afer the induction of anesthesia.
  Arms: ONDANSETRON (OS)
Drug: Droperidol — droperidol: 1.25 mg intravenous administration after the induction of anesthesia.
  Arms: DROPERIDOL (DRO)
Drug: Dexamethasone — dexametasone: 4 mg intravenous administration after the induction of anesthesia.
  Arms: DEXAMETHASONE (DEXA)

SUMMARY:
The purpose of our study is to determine if there is an antagonism between drugs used in the prevention of postoperative nausea and vomiting (PONV) on the analgesia led by acetaminophen after thyroidectomy.

DETAILED DESCRIPTION:
It was shown that there was an antagonism of the ondansetron on the analgesia led by acetaminophen in a model of nociception by electrical stimulation using the PainMatcher in healthy volunteers. Our study try to determinate if a such antagonism exist in clinical conditions : 66 patients with an Apfel-score II undergoing thyroidectomy were randomized in 3 equal groups. Each group received an antiemetic (ondansetron, droperidol or dexamethasone) at the begining of the intervention and paracetamol at the end of the intervention for the postoperative analgesia. During 2 hours in the postoperative unit, we raised : the electrical pain's threshold with the PainMatcher, the numeric pain intensity scale and the presence of nausea or vomiting. For each patients we determined the cytochrome P450 2D6 activity that should have been able to explain a diminution of ondansetron's efficiency. Paracetamol blood levels were also raised in the postoperative unit.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thyroidectomy without lymph node dissection
* American Society of Anesthesiologists physical status from I to III
* Apfel-score equal to 2
* informed consent signed

Exclusion Criteria:

* pregnant and breast-feeding women
* addictive disorders
* psychic diseases
* allergy or contra-indication to a drug used in the study
* presence of postoperative nausea or vomiting
* administration of glucocorticoid for protecting recurrent laryngeal nerve.
* protocol not respected
* protocol refused by the patient
* intellectual handicap

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
"electric nociception threshold" measured by PainMatcher | during 2 hours after thyroidectomy in the postoperative care unit
  The PainMatcher is a pain self-assessment device using the electric stimulation of the median nerve. The patient maintains a pressure on an electrode box between the thumb and the index finger, creating a current of increasing intensity. The threshold of pain sensation is obtained when the patient releases his fingers from the electrode box. So whe raise the electric nociceptive threshold showned by the PainMatcher. We realize two measures and consider the second one.
  objective measure.

SECONDARY OUTCOMES:
numeric rating scale score | during 2 hours after thyroidectomy in the postoperative care unit
  to evaluate the sensation of pain with a 11 levels going from 0 ( no pain) to 10 ( worst pain imaginable).
  subjective measure.
need in rescue analgesia with nefopam in case of numeric rating scale score > 4 | during 2 hours after thyroidectomy in the postoperative care unit
presence of postoperative nausea and vomiting | during the 2 hours after thyroidectomy in the postoperative care unit

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD,PhD, Principal Investigator — University hospital of Lille
Locations (1):
- Hôpital Claude Huriez, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905
- [Background] Girard P, Pansart Y, Coppe MC, Niedergang B, Gillardin JM. Modulation of paracetamol and nefopam antinociception by serotonin 5-HT(3) receptor antagonists in mice. Pharmacology. 2009;83(4):243-6. doi: 10.1159/000207448. Epub 2009 Mar 9. PMID 19270466
- [Background] Courade JP, Chassaing C, Bardin L, Alloui A, Eschalier A. 5-HT receptor subtypes involved in the spinal antinociceptive effect of acetaminophen in rats. Eur J Pharmacol. 2001 Nov 30;432(1):1-7. doi: 10.1016/s0014-2999(01)01464-9. PMID 11734181
- [Background] Pickering G, Esteve V, Loriot MA, Eschalier A, Dubray C. Acetaminophen reinforces descending inhibitory pain pathways. Clin Pharmacol Ther. 2008 Jul;84(1):47-51. doi: 10.1038/sj.clpt.6100403. Epub 2007 Oct 24. PMID 17957182
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] Apfel CC, Bacher A, Biedler A, Danner K, Danzeisen O, Eberhart LH, Forst H, Fritz G, Hergert M, Frings G, Goebel A, Hopf HB, Kerger H, Kranke P, Lange M, Mertzlufft F, Motsch J, Paura A, Roewer N, Schneider E, Stoecklein K, Wermelt J, Zernak C. [A factorial trial of six interventions for the prevention of postoperative nausea and vomiting]. Anaesthesist. 2005 Mar;54(3):201-9. doi: 10.1007/s00101-005-0803-8. German. PMID 15731931
- [Background] Kaiser R, Sezer O, Papies A, Bauer S, Schelenz C, Tremblay PB, Possinger K, Roots I, Brockmoller J. Patient-tailored antiemetic treatment with 5-hydroxytryptamine type 3 receptor antagonists according to cytochrome P-450 2D6 genotypes. J Clin Oncol. 2002 Jun 15;20(12):2805-11. doi: 10.1200/JCO.2002.09.064. PMID 12065557
- [Background] Nielsen M, Olsen NV. Genetic polymorphisms in the cytochrome P450 system and efficacy of 5-hydroxytryptamine type 3 receptor antagonists for postoperative nausea and vomiting. Br J Anaesth. 2008 Oct;101(4):441-5. doi: 10.1093/bja/aen246. No abstract available. PMID 18782884
- [Background] Candiotti KA, Birnbach DJ, Lubarsky DA, Nhuch F, Kamat A, Koch WH, Nikoloff M, Wu L, Andrews D. The impact of pharmacogenomics on postoperative nausea and vomiting: do CYP2D6 allele copy number and polymorphisms affect the success or failure of ondansetron prophylaxis? Anesthesiology. 2005 Mar;102(3):543-9. doi: 10.1097/00000542-200503000-00011. PMID 15731591
- [Background] Pelissier T, Alloui A, Paeile C, Eschalier A. Evidence of a central antinociceptive effect of paracetamol involving spinal 5HT3 receptors. Neuroreport. 1995 Jul 31;6(11):1546-8. doi: 10.1097/00001756-199507310-00020. PMID 7579145
- [Background] Pelissier T, Alloui A, Caussade F, Dubray C, Cloarec A, Lavarenne J, Eschalier A. Paracetamol exerts a spinal antinociceptive effect involving an indirect interaction with 5-hydroxytryptamine3 receptors: in vivo and in vitro evidence. J Pharmacol Exp Ther. 1996 Jul;278(1):8-14. PMID 8764329
- [Background] Alloui A, Chassaing C, Schmidt J, Ardid D, Dubray C, Cloarec A, Eschalier A. Paracetamol exerts a spinal, tropisetron-reversible, antinociceptive effect in an inflammatory pain model in rats. Eur J Pharmacol. 2002 May 17;443(1-3):71-7. doi: 10.1016/s0014-2999(02)01578-9. PMID 12044794
- [Background] Lund I, Lundeberg T, Kowalski J, Sandberg L, Budh CN, Svensson E. Evaluation of variations in sensory and pain threshold assessments by electrocutaneous stimulation. Physiother Theory Pract. 2005 Apr-Jun;21(2):81-92. doi: 10.1080/09593980590922307. PMID 16392461
- [Background] Nielsen PR, Norgaard L, Rasmussen LS, Kehlet H. Prediction of post-operative pain by an electrical pain stimulus. Acta Anaesthesiol Scand. 2007 May;51(5):582-6. doi: 10.1111/j.1399-6576.2007.01271.x. PMID 17430320
- [Background] Fujii Y, Nakayama M. Efficacy of dexamethasone for reducing postoperative nausea and vomiting and analgesic requirements after thyroidectomy. Otolaryngol Head Neck Surg. 2007 Feb;136(2):274-7. doi: 10.1016/j.otohns.2006.09.013. PMID 17275553
- [Background] Samer CF, Piguet V, Dayer P, Desmeules JA. [Genetic polymorphism and drug interactions: their importance in the treatment of pain]. Can J Anaesth. 2005 Oct;52(8):806-21. doi: 10.1007/BF03021775. French. PMID 16189332
- [Background] Lo Y, Chia YY, Liu K, Ko NH. Morphine sparing with droperidol in patient-controlled analgesia. J Clin Anesth. 2005 Jun;17(4):271-5. doi: 10.1016/j.jclinane.2004.08.010. PMID 15950851
- [Background] McCleane GJ, Suzuki R, Dickenson AH. Does a single intravenous injection of the 5HT3 receptor antagonist ondansetron have an analgesic effect in neuropathic pain? A double-blinded, placebo-controlled cross-over study. Anesth Analg. 2003 Nov;97(5):1474-1478. doi: 10.1213/01.ANE.0000085640.69855.51. PMID 14570668
- [Background] Andrieu G, Amrouni H, Robin E, Carnaille B, Wattier JM, Pattou F, Vallet B, Lebuffe G. Analgesic efficacy of bilateral superficial cervical plexus block administered before thyroid surgery under general anaesthesia. Br J Anaesth. 2007 Oct;99(4):561-6. doi: 10.1093/bja/aem230. Epub 2007 Aug 6. PMID 17681971